CLINICAL TRIAL: NCT01449201
Title: Phase II Trial of PF-00299804 in Patients With Metastatic/Recurrent Head and Neck Squamous Cell Carcinoma (HNSCC) After Failure of Platinum-containing Therapy
Brief Title: PF-00299804 in Patients With Head and Neck Squamous Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Byoung Chul Cho, assistant professor, Yonsei University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2011-0434
Record Dates: First submitted 2011-10-04; First posted 2011-10-10 (Estimated); Last update posted 2014-09-30 (Estimated); Status verified 2014-09

CONDITIONS: Head Neck Cancer Squamous Cell Metastatic; Head Neck Cancer Squamous Cell Recurrent
Keywords: PF-00299804, head and neck cancer, squamous cell carcinoma
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Squamous Cell | interventions — dacomitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PF-00299804 (Experimental)
  Interventions: Drug: PF-00299804

INTERVENTIONS:
Drug: PF-00299804 — 45 mg P.O. Daily (28-day treatment as one treatment cycle)

SUMMARY:
Epidermal growth factor receptor (EGFR) is often over-expressed, and have been related to poor prognosis in patients with HNSCC. EGFR targeting strategies showed clinical anti-tumor efficacy in patients with HNSCC. PF-00299804 is a second-generation quinazoline-based irreversible pan-HER inhibitor. In preclinical studies, PF-00299804 has much lower IC50 values than gefitinib in cell lines engineered to express EGFRvIII mutations (1.2 nM versus 2,700 nM) and produces tumor growth inhibition in gefitinib-resistant xenografts. A phase II trial of PF-00299804 in patients with recurrent or metastatic HNSCC is currently ongoing and preliminary report in ASCO 2010 showed its anti-tumor activity against HNSCC. The investigators suggest a phase II trial of pan-HER inhibitor PF-00299804 in patients with recurrent or metastatic HNSCC previously treated with platinum-based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed squamous cell carcinoma of head and neck
* Age ≥ 18
* ECOG PS 0-2
* Documented progressive disease after platinum-based systemic chemotherapy (either cisplatin or carboplatin) with or without cetuximab
* At least one bidimensionally measurable disease
* Adequate organ function for treatment
* Availability of tumor tissue for molecular analysis (archival or rebiopsy tissue)

Exclusion Criteria:

* Nasopharyngeal carcinoma
* Eligibility for local therapy (surgery or radiotherapy)
* Previous treatment with small molecule EGFR tyrosine kinase inhibitors
* More than one systemic chemotherapy
* Any major operation or irradiation within 4 weeks of baseline disease assessment
* Any clinically significant gastrointestinal abnormalities which may impair intake or absorption of the study drug
* CNS metastasis with continuous corticosteroid use within 4 weeks of baseline disease assessment
* Patients with known interstitial lung disease
* Patients with uncontrolled or significant cardiovascular disease (AMI within 12 months, Unstable angina within 6 months, NYHA Class III, IV Congestive heart failure or left ventricular ejection fraction below local institutional lower limit of normal or below 45%, Congenital long QT syndrome, Any significant ventricular arrhythmia, Any uncontrolled second or third degree heart block, Uncontrolled hypertension)
* Concomitant malignancy (except adequately treated basal cell cancer of skin or cervical cancer in situ)
* Pregnant or breast-feeding women
* Other severe acute or chronic medical condition or laboratory abnormality that may increase the risk associated with trial participation or investigational product administration or may interfere with the interpretation of trial results and, in the judgment of the investigator, would make the patient inappropriate for entry into this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2011-10; Primary Completion 2013-10 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Response rate | every 8 weeks
  Tumor assessment by RECIST criteria version 1.1 will be followed every 8 weeks treatment until disease progression

SECONDARY OUTCOMES:
Best objective response | every 8 weeks
  Tumor assessment by RECIST criteria version 1.1 will be followed every 8 weeks treatment until disease progression
Progression-free survival | every 8 weeks
  from C1D1 until confirmed disease progression or death
Overall survival | every 12 weeks
  from C1D1 to death
Toxicity profile | every 4 weeks
  from C1D1 to 1 months after the last dose adminitration

CONTACTS AND LOCATIONS:
Overall Officials: Byoung Chul Cho, M.D.,Ph.D., Principal Investigator — Yonsei University
Locations (6):
- South Korea (6):
  - Severance Hospital, Seoul, Seoul
  - Chilgok Kyungpook National University Hospital, Daegu
  - Dongsan Medical Center, Daegu
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital Cancer Center, Seoul